CLINICAL TRIAL: NCT06443983
Title: The Effect of Artificial Intelligence Supported Case Analysis on Nursing Students' Case Management Performance and Satisfaction: A Randomized Controlled Trial
Brief Title: Artificial Intelligence Supported Case Analysis on Nursing Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Seda Akutay, Research Assistant, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ErciyesUniversity
Record Dates: First submitted 2024-05-27; First posted 2024-06-05 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-05

CONDITIONS: Artificial Intelligence; Nursing Education; Nursing Students

STUDY DESIGN:
Intervention Model Description: In this study, students will be divided into two groups: those who take an AI-supported case lesson and those who take a standard case lesson.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI-supported case lesson group (Experimental): Students in this group will take an artificial intelligence-supported in-class case analysis lesson.
  Interventions: Other: AI-supported case
- Standard case lesson group (No Intervention): Students in this group will receive a standard in-class case lesson narrated by the instructor.

INTERVENTIONS:
Other: AI-supported case — In the artificial intelligence-supported case lesson, students will listen to audio and visual content prepared by artificial intelligence.
  Arms: AI-supported case lesson group

SUMMARY:
Background: Rapid developments in the field of artificial intelligence have begun to necessitate changes and transformations in nursing education.

Objective: This study aimed to evaluate the impact of an artificial intelligence-supported case created in the in-class case analysis lecture for nursing students on students' case management performance and satisfaction.

Design: This study was a randomized controlled trial. Method: The study involved 188 third-year nursing students who were randomly assigned to either the AI group (n=94) and control group (n=94). An information form, case evaluation form, knowledge test, and Mentimeter application were used to assess the students' case management performance and nursing diagnoses. The level of satisfaction with the case analysis lecture was evaluated using the VAS scale.

ELIGIBILITY:
Inclusion Criteria:

* having taken nursing process lecture before
* having planned care for at least one surgical patient in clinical practice before
* having a mobile phone with internet connection

Exclusion Criteria:

* not attending the case analysis lecture
* not being an active student
* incomplete completion of the data collection forms
* not accepting to participate in the study

Ages: 20 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 188 (Actual)
Dates: Start 2024-02-27 (Actual); Primary Completion 2024-03-27 (Actual); Study Completion 2024-03-27 (Actual)

PRIMARY OUTCOMES:
Case management performance | 3 hours
  The performances of all students included in this study regarding the case lesson were evaluated by means of a knowledge test consisting of 10 questions and a Mentimeter application in which they could indicate their nursing diagnoses. The students will solve the tests after the case lessons are completed. The scores that can be obtained from the tests are between 0-100. As the score of the students increases, it can be interpreted that the level of knowledge increases. In the Mentimeter application, students will be asked to write 5 nursing diagnoses. There is no scoring here, but the application creates a word cloud with the most given answer in a larger font size.
Case Satisfaction | 3 hours
  The level of satisfaction with the case analysis lecture was evaluated using the VAS scale. The VAS scale is scored between 1-10. Students indicate their satisfaction with the processing of the case lesson. High scores on the VAS indicate a high level of satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Seda Akutay, Ress. Asst., Principal Investigator — TC Erciyes University
Locations (1):
- Erciyes University, Kayseri, Turkey (Türkiye)

REFERENCES:
- [Derived] Akutay S, Yuceler Kacmaz H, Kahraman H. The effect of artificial intelligence supported case analysis on nursing students' case management performance and satisfaction: A randomized controlled trial. Nurse Educ Pract. 2024 Oct;80:104142. doi: 10.1016/j.nepr.2024.104142. Epub 2024 Sep 12. PMID 39299058